CLINICAL TRIAL: NCT01791101
Title: Eltrombopag in Patients With Delayed Post Transplant Thrombocytopenia.
Acronym: ITP0511
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITP0511; 2011-004608-39 (EudraCT Number)
Record Dates: First submitted 2013-02-12; First posted 2013-02-13 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Thrombocytopenia
Keywords: Thrombocytopenia; Eltrombopag
MeSH Terms: conditions — Thrombocytopenia | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eltrombopag (Experimental): Eltrombopag 50 mg/daily.
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag

SUMMARY:
This is a Phase II multicentre study. Patients will be administered eltrombopag 50 mg/daily. If patients don't achieve response after 2 months of therapy they will stop eltrombopag; if patients will achieve response after 2 months of therapy, they will continue eltrombopag for a maximum period of 24 months; 40 patients are needed. In stage I, 22 patients will be enrolled; if ≤ 4 responses at the first evaluation after 2 months (18%) will be seen, the trial will be stopped; if 5 or more responses will be seen, the accrual will continue. In stage II, 18 more patients will be enrolled. If ≤ 12 (30%) responses will be observed out of 40 patients, it will be concluded that the study drug is not active enough. If ≥ 13 responses will be observed, it will be concluded that eltrombopag is worth of further studies.

DETAILED DESCRIPTION:
The incidence of delayed thrombocytopenia in patients who undergo allogeneic hemopoietic stem cell transplant (SCT) is nearly 20-40% (1-2). Chronic graft versus host disease (cGVHD) seems to be the most frequent pathologic condition associated with post SCT delayed thrombocytopenia. Previous studies indicated the occurrence of delayed thrombocytopenia as a poor prognostic factor for the outcome of patients undergoing SCT, particularly for those patients with cGVHD. In our experience, 27 out of 71 patients (38%) developed post SCT delayed thrombocytopenia, with a median platelet count of 29 x 109/L (range 7-86 x 109/L); cGVHD was associated with delayed thrombocytopenia in 54% of cases. The platelet count was >50 <100 x 109/L in 8 patients (30%) patients and 50 x 109/L in 19 (70%) among whom 9 had 20 x 109/L. The median post SCT survival was 12 months in patients who developed delayed thrombocytopenia vs. > 36 months in patients without delayed thrombocytopenia. The rate of patients alive 12, 24 and 33 months after SCT was 41%, 41% and 7% among patients with delayed thrombocytopenia vs. 93%, 87% and 87% (p< 0.0001). In patients with cGVHD the incidence of mortality was significantly higher in those who developed post SCT thrombocytopenia, i.e. 8 out of 13 (61.5%) vs. 2 out of 19 (10.5%) (p=0.005). Our data confirms the results of previous studies. Therefore, the occurrence of delayed thrombocytopenia in patients undergoing SCT is a very poor prognostic factor and the improvement of this condition may favourably affect patients' outcome. The pathophysiology of cGVHD relayed post SCT delayed thrombocytopenia is complex and only partial understood. Biological and clinical evidences support an autoimmune-like thrombocytopenia with increased platelet destruction; this mechanism is also suggested by the response to some therapeutic strategies generally adopted to treat classical immune thrombocytopenia as steroids, high dose intravenous immunoglobulin, splenectomy, rituximab. However a mechanism consistent with impaired platelet production has also been suggested. Adopting an index for plasma glycocalicin, plasma thrombopoietin (TPO), and circulating B cells producing anti-GPIIb-IIIa antibodies, Yamazaki et al. studied 23 SCT recipients who had prolonged and isolated thrombocytopenia with no apparent causes such as engraftment failure, recurrence of the underlying malignancy, microangiopathy or drugs and compared data with those observed in a similar cohort of SCT recipients with no thrombocytopenia, in patients with primary immune thrombocytopenia (ITP) and aplastic anemia. Despite the frequent occurrence of an antiplatelet antibody response, patients with post SCT thrombocytopenia showed a glycocalicin index and TPO status similar to that seen in aplastic anemia. TPO levels were normal in nearly 30% of patients. Recently, Bao et al. showed an improved regulatory T-cell (T-regs) activity in patients with chronic primary immune thrombocytopenia (ITP) treated with thrombolytic agents, suggesting a possible role of platelet count in improving T-reg function and restore immune tolerance.

On this grounds and similarly to ITP, the stimulation of thrombopoiesis with the thrombolytic agents could be beneficial in some patients with persistent post SCT thrombocytopenia both on platelet count and on cGVHD manifestations. Eltrombopag (Revolade) is a thrombopoietin receptor agonist indicated for the treatment of adult patients with ITP relapsed/refractory to splenectomy; eltrombopag may be considered as second line treatment for adult non-splenectomised patients where surgery is contraindicated. Eltrombopag is also under development for the treatment of thrombocytopenia due to hepatitis C virus HCV, for chemotherapy-induced thrombocytopenia and in MDS/AML.

ELIGIBILITY:
Inclusion Criteria:

* Patients develop delayed thrombocytopenia, i.e. Platelet count 50 x 109/l 3 months after SCT;
* Patients underwent allogeneic SCT with match related or unrelated donor;
* Patients develop CGVHD-related delayed thrombocytopenia. The definition of cGVHD-related delayed thrombocytopenia is: platelet count 50 x 109/l from month 3 from SCT and presence of any clinical, radiological and/or laboratory finding indicative of cGVHD (all grades); - Patients underwent SCT because of lymphoma (Hodgkin or non-Hodgkin, indolent or aggressive), or multiple myeloma;
* Sexually active males who accept to use a condom during intercourse while taking the drug and for 12 months after stopping treatment as they should not father a child in this period. A condom is required to be used also by vasectomised men (as well as during intercourse with a male partner) in order to prevent delivery of the drug via seminal fluid. Refer also to Appendix C. Female subjects of non-childbearing potential may be enrolled in the study; For this study population, non-childbearing potential is defined as current tubal ligation, hysterectomy, ovariectomy or post-menopause (please refer to Appendix C);
* OR Female subjects of childbearing potential may be enrolled in the study, if the subject has practiced adequate contraception for 30 days prior to start of eltrombopag, has a negative pregnancy test prior to start of eltrombopag, and has agreed to continue adequate contraception during the entire treatment period and for 6 months after completion of the treatment.
* Written informed consent obtained from the subject.

Exclusion Criteria:

* Patients underwent SCT with aplo-identical donor or cord blood;
* Patients underwent SCT for diseases different from lymphoma or multiple myeloma;
* Patients have life threatening bleeding complications;
* Patients have an expected survival < 1 month;
* Patients have delayed thrombocytopenia related to medical conditions other then cGVHD;
* Patients have progressive non stabilized cGVHD necessitating intensification of immune suppressive treatment in the last 2 weeks;
* Patients need to introduce or increase the dosage of steroids, any other immune suppressive or cytotoxic agent at the time of enrolment into the study or start of eltrombopag; patients already in treatment with a fixed, stabilized dosage of steroids or other immune suppressive agents because of cGVHD may be included into the study;
* Patients received concomitant erythropoietin treatment; Patients have active deep venous thrombosis (DVT);
* Patients have venous occlusive disease (VOD);
* Patients have grade 3-4 hyper bilirubinemia; elevation of hepatic enzymes because of cGVHD should not be considered criteria of exclusion.
* Patients with baseline elevation of hepatic enzymes will be monitored carefully in order to point out possible addictive eltrombopag- related hepatotoxicity;
* Patients have hepatic cirrhosis;
* Patients have transplant related-microangiopathy;
* Patients have active infections (CMV reactivation included);
* Patients have hypersensitive to study drug;
* Patients are unable to stop medications that are known to cause a drug-drug interaction with eltrombopag.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-09-16 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Number of patients who achieve both a platelet count ≥ 50 x 109/L and have doubled their baseline platelet count. | Two months after treatment with eltrombopag.
  Response rate (OR), i.e. the number of patients who achieve both a platelet count ≥ 50 x 109/L and have doubled their baseline platelet count, two months after treatment with eltrombopag. The primary endpoint will be considered for all the treated population according to the intention-to-treat and in the evaluable population, i.e. all patients treated with eltrombopag for at least 3 weeks or who interrupted eltrombopag because of toxic events. A transient increase of platelet count after the administration of iv immunoglobulin given for anti- microbial purpose will not be considered criteria of response.

SECONDARY OUTCOMES:
Number of adverse events. | After 4 years from study entry.
  Safety profile Incidence of AEs according to NCI Common Terminology Criteria for Adverse Events v 4.0 [NCI CTCAE] toxicity scale.
Number of surviving patients. | At 4 years from study entry.
  Overall Survival OS will be evaluated with Kaplan Meyer and compared with historical patients who developed post SCT delayed thrombocytopenia.
Number of bleeding events. | After 4 years from study entry.
  Bleeding events Bleeding events will be evaluated according to the WHO bleeding scale (grade 0, no bleeding; grade 1, petechiae; grade 2, mild blood loss; grade 3, gross blood loss; grade 4, debilitating blood loss).
Characteristics of TPO serum level. | After 4 years from study entry.
  TPO serum level TPO will be measured using a Human TPO duo-set assay (R&D System). This assay employs the quantitative sandwich enzyme immunoassay technique to evaluate the concentration of TPO in plasma or serum.
Patients T-reg activity. | After 4 years from study entry.
  T-reg activity T-reg activity will be evaluated by flow cytometric analysis of CD4+ CD25+ FOXP3+ lymphocytes in a mixed lymphocyte population.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Zaja, Principal Investigator — Clinica Ematologica, DISM, Azienda Ospedaliera Universitaria S. M. Misericordia
Locations (16):
- Italy (16):
  - UO Ematologia con trapianto-Università degli Studi di Bari Aldo Moro, Bari
  - Divisione di Ematologia - Ospedali Riuniti, Bergamo
  - USD Trapianti di midollo per adulti - Cattedra di Ematologia - Università degli Studi di Brescia, Brescia
  - Ospedale Santa Croce Divisione di Ematologia Cuneo, Catania
  - Ospedale Santa Croce Divisione di Ematologia Cuneo, Cuneo
  - Policlinico di Careggi, Florence
  - Divisione Ematologia 2 - Azienda Ospedaliera Universitaria - S.Martino, Genova
  - Unità Trapianto di Midollo Ist. Nazionale Tumori, Milan
  - La Maddalena Casa di Cura di Alta Specialità Dipartimento Oncologico di III Livello, Palermo
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - Università degli Studi - Policlinico di Tor Vergata, Roma
  - Clinica Ematologica - Policlinico Universitario, Udine
  - ULSS N. 6 Ospedale S. Bortolo, Vicenza
  - ULSS N.6 Osp. S. Bortolo, Vicenza

IPD SHARING:
Plan to Share IPD: No